CLINICAL TRIAL: NCT04148157
Title: Prospective, Observational Study of the Factors Affecting Patient and Physician Perceptions of Quality of Life in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Quality of Life in IPF - Patient and Physician Perceptions
Acronym: QUALY-IPF-PPP
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Washington Research Foundation (Unknown)
Responsible Party: Principal Investigator, Ganesh Raghu, Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00008283
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Quality of Life; Questionnaire
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the differences between patient's and their physicians' perception of quality of life and the effect of disease severity and co-morbidities. Patients and physicians will complete two sets of questionnaires at an initial clinic visit and again six months later.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis is a progressive and debilitating disease characterized by progressive scarring of the lung parenchyma of unknown cause. In the US approximately 100,000 individuals have been diagnosed with this disease and the only cure available is lung transplantation. There have been two drugs approved by the FDA for treatment of IPF which have demonstrated the ability to slow disease progression but have no impact on quality of life.

Symptoms of IPF include shortness of breath, cough, and fatigue which all contribute to a decreased quality of life. Additionally, these symptoms and the need for supplemental oxygen use causes significant psychological and social impairment. Multiple questionnaires have been used to measure patient reported quality of life in both clinical and research settings. The King's Brief Interstitial Lung Disease (KBILD) Questionnaire is a disease-specific patient reported outcome measure and has been validated across several different patient groups and countries. Additionally, the EuroQol group has developed the EuroQol five dimensional 5-Level (EQ-5D-5L) questionnaire which is a non-disease specific assessment of health-related quality of life and has not yet been widely used in a population of patients with IPF.

Significant disparity between patient and physician perception of quality of life has been demonstrated across different disease processes. While there are many contributing factors to overall wellbeing the general assumption is that with more advanced disease quality of life predictably decreases. The investigators plan to test this hypothesis to better understand the complex relationship between chronic disease and quality of life in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a multidisciplinary diagnosis of IPF according to the 2018 ATS/ERS/JRS/ALAT Clinical Practice Guidelines.
* All ranges of disease severity based on pulmonary function testing: forced vital capacity (FVC) and diffusing capacity (DLCO).

Exclusion Criteria:

* Any impairment or co-morbid disease that results in an inability to read or understand a questionnaire or provide informed consent. The study team member will make this determination according to their best clinical judgement.
* The questionnaires will be administered in English language only and thus this study will be conducted in patients who are able to read, write, and speak English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in this study will hold a diagnosis of Idiopathic Pulmonary Fibrosis (IPF) as detailed above. As IPF occurs only in adults all subjects must be 18 years of age or older. Both men and women will be recruited for the study. Subjects of all ethnicities and racial minorities will be recruited. Physicians who are seeing these patients for regular clinical visits during the study will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Patient and Physician Responses to the Kings Brief ILD (K-BILD) Questionnaire | 6 months
  A comparison of physician and patient reported quality of life based on responses to the Kings Brief ILD Questionnaire (K-BILD). The domain and total score ranges are 0-100 where a score of 100 represents best health status.
Patient and Physician Responses to the EuroQol five dimensional 5-Level (EQ-5D-5L) questionnaire | 6 months
  A comparison of physician and patient reported quality of life based on responses to the EuroQol five dimensional 5-Level (EQ-5D-5L) questionnaire. The domain ranges are 1-5 and the total score ranges are 5-25 where a score of 5 represents best health status. The visual analog scale portion of the questionnaire ranges from 0 to 100 where a score of 100 represents best health status.
Patient and Physician Responses to the Raghu Quality of Life in Interstitial Lung Disease (RQ-LIFE-ILD) Questionnaire | 6 months
  A comparison of physician and patient reported quality of life based on responses to a novel visual analog scale questionnaire the Raghu Quality of Life in Interstitial Lung Disease (RQ-LIFE-ILD) Questionnaire. The domain ranges are 0 to 10 and the total score ranges are 0 to 50 where a score of 0 represents best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Raghu, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington - Center for Interstitial Lung Disease, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scallan C, Strand L, Hayes J, Kadura S, Collins B, Ho L, Spada C, Canestaro W, Kolb M, Raghu G. R-scale for pulmonary fibrosis: a simple, visual tool for the assessment of health-related quality of life. Eur Respir J. 2022 Jan 13;59(1):2100917. doi: 10.1183/13993003.00917-2021. Print 2022 Jan. PMID 34112729